CLINICAL TRIAL: NCT01946581
Title: Retrospective Patient Satisfaction Survey in Subjects With Tecnis Intra Ocular Lenses Cataracts Surgery
Brief Title: Retrospective Patient Satisfaction Survey in Subjects With Tecnis Intra Ocular Lenses and Cataracts Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MDbackline, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: JH SAT 2013
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cataract Surgery
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery

SUMMARY:
Define what factors correlate with higher degrees of patient satisfaction and dissatisfaction among patients who have recently undergone cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated bilateral cataract surgery with a Tecnis Multifocal or monofocal implant completed at least 60 days before the survey date.
* Patient with and without astigmatic keratotomy will be included.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.)
* Patients with ≥ grade 1 posterior capsule opacity at their last visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have had Cataract Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Patient overall satisfaction post Cataract surgery | 60 plus days Post surgery
  Patient will be given a satisfaction survey based on overall satisfaction:
  * Motivations for choosing their surgeon and for selecting an IOL choice
  * Fears that they had before surgery
  * Degree of spectacle independence for activities, including driving (day and night), watching television, computer use, reading print material, using their mobile phone
  * Degree of overall satisfaction with vision
  * Degree to which they notice unexpected side effects (dysphotopsias)
  * Degree to which they felt informed about any side effects they did experience
  * Activities for which they would like to see better
  * Willingness to refer friends for the same surgery
  * Whether they have already referred friends for the same surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — MD backline; John Hovanesian, MD, Study Director — MD Backline
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States